CLINICAL TRIAL: NCT06291818
Title: Self-Adhering Magnetic Device to Treat Corneal Exposure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Peter Setabutr, Director, Oculoplastic & Reconstructive Surgery Service Director, Millennium Park Eye Center, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-0917
Record Dates: First submitted 2024-01-26; First posted 2024-03-04 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Paralytic Lagophthalmos; Corneal Exposure
MeSH Terms: conditions — Lagophthalmos

STUDY DESIGN:
Intervention Model Description: temporary magnetic system for tarsorrhaphy (MST)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assess the performance of this novel eyelid closure device in vivo (Other): The primary goal of this study is to determine the feasibility and success of a temporary magnetic system for tarsorrhaphy (MST) to provide adequate closure of the eyes for ultimate use in conditions causing lagophthalmos (a disorder in eyelid closure). In this disorder, people are unable to sufficiently cover their cornea (the front of the eye), which can lead to dryness, infection, scarring and even blindness. Current therapies are invasive, involving local anesthesia and surgeries, and have a negative cosmetic impact.
  Interventions: Device: temporary magnetic system for tarsorrhaphy (MST)

INTERVENTIONS:
Device: temporary magnetic system for tarsorrhaphy (MST) — cutting-edge technology has produced smaller magnets with stronger magnetic fields, prompting experts to revisit the use of magnets to facilitate eyelid closure

SUMMARY:
Paralytic lagophthalmos can be difficult to treat and manage. It has a host of causes and effects, one of which (for the latter) is exposure keratopathy. Untreated, this can lead to corneal ulceration, inflammation, and potentially blindness. Despite a variety of attempts at treating this complex condition, none have satisfactorily reduced complications ranging from ease of use to aesthetics. With improvement in magnetic technology, however, that may change. Barmettler et al (2014) have demonstrated preliminary success of externally affixed magnets in closing both model and patient eyelids. As such, we hypothesize that magnetic devices can be used to treat corneal exposure by controlling eyelid position.

DETAILED DESCRIPTION:
Patients who suffer from lagophthalmos cannot close their eyelids completely. In paralytic lagophthalmos, this physical incapability is caused by paralysis of the seventh cranial nerve. Causes of this paralysis include Bell's palsy, vascular accidents, injury, trauma, and tumors. Complications can include irritation, ulceration, and perforation of the cornea; exposure and neurotrophic keratopathy; persistent epithelial defects; and potential blindness.

Due to the myriad causes and complications, management of paralytic lagophthalmos has proven difficult, and existing methods of treatment each have shortcomings. Initial, mainly conservative, and supportive, management includes use of ocular lubricants, moisture chambers, eyelid taping, adhesive eyelid weights, bandage contact lenses, botulinum toxin, and hyaluronic-acid gel fillers. Ephemeral benefits and low patient compliance due to frequency of application often leave these treatments destined for failure.

As such, surgical intervention is subsequently necessary, although surgical methods have been shown to be flawed as well. Tarsorrhaphies are static surgical procedures in which the eyelids are partially or completely sewn together to narrow the palpebral fissure. Although effective in healing corneal lesions preventing excessive corneal exposure, tarsorrhaphies often require repeated suturing, which both increases inflammatory response of the eyelids to the sutures and, much to patients' discontent, decreases cosmesis. Loosening of the sutures, restricted peripheral vision, and trichiasis are additional potential negative outcomes. In another static procedure known as "lid loading", gold or platinum weights are implanted into the eyelid. However, these are susceptible to extrusion and can cause blepharoptosis (drooping of the upper eyelid), allergic reactions, and-when the patient is supine-incomplete eyelid closure. Cartilage grafts as weights fail to treat severe cases of paralytic lagophthalmos. Palpebral springs, used in a dynamic procedure, require numerous revisions and are thus impractical for long-term benefits.

Certain clinical situations may develop into paralytic lagophthalmos and cause downstream effects later on. These clinical conditions include corneal abrasions, or scratches of the cornea, as well as a surgical procedure called eye enucleation, or the surgical removal of the eye for other reasons (typically but not always replaced with a glass or prosthetic eye). Because these conditions or procedures may be associated with paralytic lagophthalmos, improving eyelid closure before development of permanent lagophthalmos may be critical in preventing future corneal ulcers and worse conditions of the eye.

In addition to conservative and surgical approaches to management of paralytic lagophthalmos and the resulting exposure keratopathy, clinicians and researchers have also utilized magnets for eyelid closure. First suggested in 1957, this method grew in favor in the decades to follow, as several major studies were published indicating its success in both cosmetics and functionality. However, due to limited technology and moderate amount of magnet extrusion, this method was temporarily abandoned. Today, cutting-edge technology has produced smaller magnets with stronger magnetic fields, prompting experts to revisit the use of magnets to facilitate eyelid closure. In a study conducted by Barmettler magnets embedded in biocompatible molds were affixed in two configurations: 1) to the upper and lower eyelids, or 2) to the upper eyelid and to the lower rim of the frame of a pair of eyeglasses. Initial model and patient testing were promising, but questions remain regarding the strength of magnets in disease states, size of the silicone mold, and implantability as opposed to external affixation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-80 years old.
* Patients with recent corneal abrasion and no signs of infection in the examination
* Patients with lagophthalmos
* Normal Controls

Exclusion Criteria:

* Individuals with adhesive or tape allergies.
* Individuals with a history of metal pieces/shavings embedded in the eye (such as from welding or metalworking)
* Individuals with eye infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with success of a temporary magnetic system for tarsorrhaphy | through study completion, an average of 3 years
  Use of a temporary magnetic system for tarsorrhaphy (MST) to provide adequate closure of the eyes for ultimate use in conditions causing lagophthalmos (a disorder in eyelid closure)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois - Specialty Care Building, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided